CLINICAL TRIAL: NCT06168175
Title: A Feasibility Single-center, Randomized, Double-blind, Placebo-controlled Study to Assess the Feasibility of Conducting a Full-scale Randomized Controlled Trial (RCT) Assessing Efficacy of Lactate as Adjunctive Therapy in Hospitalized Patients With Major Depressive Disorder
Brief Title: Feasibility of Conducting a Clinical Trial Assessing Efficacy of Lactate as Adjunctive Therapy in Patients With Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Fondation de Préfargier (Unknown)
Responsible Party: Principal Investigator, Sylfa Fassassi, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lac-MDD; 2023-01702 (Other: CER-VD)
Record Dates: First submitted 2023-11-10; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
Keywords: Sodium lactate; Depression; Antidepressant; Lactate
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sodium Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactate (Experimental)
  Interventions: Drug: Sodium lactate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium lactate — 2 mmol/kg, intravenous, daily for 5 consecutive days
  Arms: Lactate
Drug: Placebo — intravenous, daily for 5 consecutive days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the efficacy of lactate (a natural substance) in combination with standard antidepressant treatment, in patients hospitalized for a major depressive episode.

The main question[s] it aims to answer are:

* does lactate diminishes depression severity when administered in combination with antidepressant ?
* is it feasible to test lactate treatment in a large-scale clinical trial ? Participants will receive lactate intravenously daily (20 min infusion) for 5 days during hospitalisation (together with the standard antidepressant treatment).

Researchers will compare with a group receiving a placebo instead of lactate to see if lactate has antidepressant effects.

DETAILED DESCRIPTION:
In case of major depressive disorder (MDD), antidepressant medications are prescribed as standard treatment. The commonly used antidepressants have a delayed onset of therapeutic actions, many side effects and limited efficacy. In this regard, about 30-50% of MDD patients are unresponsive to any currently approved pharmacological treatment, emphasizing the need for novel types of drugs to treat major depression.

Several animal studies have shown that lactate, a substance naturally present in the body, has antidepressant effects.

The aim of this single-center study is to evaluate the feasibility of conducting a future large-scale clinical trial testing the efficacy of "sodium lactate" as an adjunctive treatment to a standardly prescribed antidepressant.

The study is recruiting patients hospitalized for a major depressive episode. Participants are assigned randomly to the "sodium lactate" group or the "placebo" group. The study treatment will be administered intravenously daily (2mmol/kg) for 5 days during hospitalization, in addition to standard antidepressant treatment. Patients will be followed during hospitalization and then on an outpatient basis at 6 and 12 weeks. The therapeutic effect of sodium lactate will be assessed with the MADRS score (depression severity scale) at 1, 2, 3, 6 and 12 weeks. Recruitment, adherence, retention, data completion and blinding maintenance rates will also be assessed to evaluate the feasibility. The effect on anxiety, perceived stress, insomnia, short-term depression remission rate, blood lactate level and length of hospitalization will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Study consent signed
* 18 ≤ age ≤ 65 years old
* Fluent in french
* Recently (no more than 1 week) hospitalized for a primary diagnosis of MDD
* Current major depressive episode as defined by DSM-5
* Current MADRS score ≥18
* Total number of MDD acute episodes ≤ 3
* Total number of psychiatric medications ≤ 3 at admission
* Total number of any medication ≤ 4 at admission
* No signs or evidence indicating difficult intravenous access
* Willing to hold a peripheral blood catheter for 5 days

Exclusion Criteria:

* Bipolar depression
* History of panic attacks
* Severe substance use disorders according to DSM-5-TR criteria
* Conditions predisposing to hypernatremia such as:

  * adrenocortical insufficiency,
  * diabetes type 1 and insulin-dependent type 2
  * extensive tissue injury
* Known severe renal insufficiency
* Known hepatic insufficiency (impaired lactate metabolism)
* Known history of heart failure
* Known history of Chronnic Obstructive Pulmonary Disease or respiratory failure
* Known hypersentitivity to lactate
* Hypernatremia with Na+ > 150 mmol/L (confirmed on 2 blood withdrawals)
* Blood osmolality > 320 mmol/kg H2O
* Hyperlactatemia > 2 mmol/l
* Pregnant or lactating
* Forbiden medications : Lithium
* Participation to other clinical trials
* Any medical conditions that could jeopardize patient's health in case of study participation according to the investigator
* Inability to give informed consent (without capacity for discernment) as evaluated by the psychiatrist investigator or by by a delegated physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by the recruitment rate | 12 weeks
  % of patients eligible among the informed patients
Feasibility as assessed by the adherence rate | 12 weeks
  % of patients completing the study intervention period among randomized patients
Feasibility as assessed by the retention rate | 12 weeks
  % of drop-outs among randomized patients at 3 weeks, 6 weeks and 12 weeks
Feasibility as assessed by the data completion rate of the therapeutic effect measures | 12 weeks
  % of patients with completed Montgomery Asberg Depression Rating Scale (MADRS) questionnaire at 1, 2, 3, 6 and 12 weeks among randomized patients
Feasibility as assessed by estimates of the therapeutic effect size on Montgomery Asberg Depression Rating Scale (MADRS) score | 12 weeks
  Estimate of mean difference on the change in MADRS score from baseline to week 1, 2, 3, 6 and 12 between patients randomized in lactate arm and in placebo arm, as well as their associated standard deviation.
Feasibility as assessed by the blinding maintenance rate | 12 weeks
  % of patients with sustained blinding at week 1, 2, 3, 6 and 12

SECONDARY OUTCOMES:
Anxiety | 12 weeks
  Generalized Anxiety Disorder - 7 items (GAD-7 score) ; minimum and maximum values : 0 - 21 ; Lower scores mean a better outcome
Perceived stress | 12 weeks
  Perceived Stress Scale (PSS score) ; minimum and maximum values : 0 - 40 ; Lower scores mean a better outcome
Insomnia | 12 weeks
  Insomnia Severity Index (ISI score) ; minimum and maximum values : 0 - 28 ; Lower scores mean a better outcome
Short term depression remission rate | 12 weeks
  Montgomery Asberg Depression Rating Scale (MADRS score < 7) ; minimum and maximum values : 0 - 60 ; Lower scores mean a better outcome
Hospitalization duration | 12 weeks
  Number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Marquet, MD, Study Chair — Centre Hospitalier Universitaire Vaudois